CLINICAL TRIAL: NCT04086940
Title: Lecturer of Anesthesia
Brief Title: Role of Intraoperative Beta Blocker for Morbid Obese Patients Undergoing Laparoscopic Bariatric Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, RAMY AHMED, lecturer of anesthesia at faculty of medicine ain shams university, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Ain Shams university 1
Record Dates: First submitted 2019-09-05; First posted 2019-09-12 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Intraoperative Awareness; Postoperative Pain
Keywords: role; INTRAOPERATIVE; beta blocker; bariatric surgery; morbid obese
MeSH Terms: conditions — Intraoperative Awareness; Pain, Postoperative | interventions — esmolol; Saline Solution

STUDY DESIGN:
Intervention Model Description: prospective randomized controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- esmolol(breviblock) group (Active Comparator): Patients in group E received a loading dose of esmolol(breviblock) 1 mg/kg in 50 ml isotonic saline over 30 minutes before induction of anesthesia, then followed by an infusion of esmolol 10 µg/kg/min until the end of the surgery.
  Interventions: Drug: Esmolol
- non esmolol group (Active Comparator): Patients in group N received 50 ml of isotonic saline over 30 min, followed by an infusion of isotonic saline at same rate of group E till the end of the surgery.
  Interventions: Drug: Esmolol

INTERVENTIONS:
Drug: Esmolol — preventive
  Other Names: normal saline

SUMMARY:
Using esmolol during anesthetic maintenance of laparoscopic bariatric surgery significantly decreases anesthetic, analgesic requirements, postoperative pain, PNV and postoperative hypoxia.

DETAILED DESCRIPTION:
Postoperative pain, nausea, vomiting (PNV) and hypoxia are common in relation to laparoscopic bariatric surgery. Sympatholytic drugs might decrease the need for intravenous or Inhalation anesthetics and opioids. In this study we wanted to analyze effects of esmolol on intraoperative anesthetic-analgesic requirements, postoperative analgesic requirements, postoperative pain, PNV and hypoxia.

Methods: Sixty patients have been included. Propofol, fentanyl and rocuronium were used for induction. Study groups were as follows; group E Esmolol infusion was added to maintenance anesthetics (Sevoflurane and fentanyl), group N only Sevoflurane and fentanyl was used during maintenance. They have been monitored during the intraoperative period and postoperatively for 24 h for analgesic requirements and PNV. Visual analog scale (VAS) scores for pain was also been assessed.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) I - II patients
* age between 18-59 years
* both genders
* body mass index (BMI) > 45 kg/m2

Exclusion Criteria:

* Patients with -hepatic
* renal
* cardiac
* respiratory diseases
* patients with a history of drug abuse or who were dependent on opioid drugs.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
intraoperative analgesic requirements | 6 months
  amount of narcotics and anesthetics needed
postoperative analgesic requirements | 6 months
  amount of narcotics needed

CONTACTS AND LOCATIONS:
Locations (1):
- Ramymahrose, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
after publication